CLINICAL TRIAL: NCT03988855
Title: An Exploratory, Open-Label, Oligo-Center Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Intravenous DNV3837 in Subjects With Clostridium Difficile Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deinove (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 001C16
Record Dates: First submitted 2019-06-12; First posted 2019-06-18 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Clostridium Difficile (C. Difficile)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): 10 subjects of either sex with severe or non-severe CDI will be enrolled to receive DNV3837. Treatment infusions will be administered at a constant rate resulting in a total IV infusion duration of 6 hours per day, for a total daily dose of 1.5 mg/kg actual body weight(BW)/day DNV3837. Infusions will be administered once daily for 10 consecutive days.
  Interventions: Drug: DNV3837
- Part 2 (Experimental): 30 subjects with severe or non-severe CDI will be enrolled to receive DNV3837. Treatment infusions will be administered at a constant rate resulting in a total IV infusion duration of 6 hours per day, for a total daily dose of 1.5 mg/kg actual body weight(BW)/day DNV3837. Infusions will be administered once daily for 10 consecutive days
  Interventions: Drug: DNV3837

INTERVENTIONS:
Drug: DNV3837 — Treatment infusions will be administered at a constant rate resulting in a total IV infusion duration of 6 hours per day, for a total maximum daily dose of 120 mg DNV3837. Infusions will be administered once daily for 10 consecutive days.

SUMMARY:
This is an open-label study to evaluate the safety, efficacy, and PK of DNV3837 at a dose of 1.5 mg/kg actual body weight(BW)/day administered via IV infusion in subjects with CDI. The study will be conducted in 2 subsequent parts.

In Part 1 of the study, 10 subjects of either sex with severe or non-severe CDI will be enrolled to receive DNV3837.

In Part 2 of the study, up to 30 subjects with severe or non-severe CDI will be enrolled to receive DNV3837.

In both parts of the study, treatment infusions will be administered at a constant rate resulting in a total IV infusion duration of 6 hours per day, for a total maximum daily dose of 120 mg DNV3837. Infusions will be administered once daily for 10 consecutive days. The objectives of the study are:

* To evaluate the safety of intravenous (IV) DNV3837;
* To evaluate the efficacy of IV DNV3837;
* To assess the pharmacokinetics (PK) of DNV3837 and DNV3681 in plasma and of DNV3681 in urine and feces;
* To assess C. difficile using microbiological assessments;
* To assess the proportion of subjects colonized with vancomycin-resistant enterococci (VRE), extended-spectrum beta-lactamase (ESBL) organisms, or carbapenem-resistant Enterobacteriaceae (CRE) in feces; and
* To assess changes in the fecal microbiome using 16S ribosomal ribonucleic acid (RNA) analysis

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be enrolled in the study:

1. The subject or a legally authorized representative must sign informed consent;
2. The subject must be 18 years of age;
3. Subjects must have a diagnosis of CDI defined as follows:

   1. Diarrhea, defined as a change in bowel habits, with > 3 liquid stools or unformed bowel movements (UBMs) [Bristol Stool Scale 6 or 7] or > 200 mL unformed stool for subjects having rectal collection devices in the 24 hours prior to start of study drug; AND
   2. The subject has the following positive tests on a stool sample produced within 72 hours prior to the start of study drug as determined by:

      * A positive C. difficile glutamate dehydrogenase (GDH) test by a Food and Drug Administration (FDA)-cleared enzyme immunoassay (EIA); AND
      * A positive toxin test (presence of either C. difficile Toxin A [TcdA] and/or C. difficile Toxin B [TcdB]) by an FDA-cleared EIA; OR
      * A positive toxin gene test (presence of either C. difficile Toxin A gene [tcdA] and/or C. difficile Toxin B gene [tcdB]) by an FDA-cleared nucleic acid amplification test; OR
      * A positive cell cytotoxicity neutralization assay; OR
      * positive toxigenic culture;
4. Subjects with a first episode or recurrence of CDI with at least 1 of the following criteria:

   1. Current diagnosis of non-severe CDI must have a white blood cell (WBC) count ≤15,000 cells/µL (15 × 10^9 cells/L) and serum creatinine <1.5 mg/dL;
   2. Subjects with a current diagnosis of severe CDI must have any of the following criteria:

      * WBC count >15,000 cells/µL (15 x 10^9 cells/L);
      * Serum creatinine ≥ 1.5 mg/dL;
      * Colitis on computed tomography or magnetic resonance imaging scan or ultrasound; OR
      * Severe abdominal pain, vomiting, ileus, temperature >38.9°C, or albumin level <2.5 g/dL in which CDI is strongly suspected and other non-CDI causes of infection have been ruled out;
   3. Is currently failing antibiotic therapy for CDI, as defined by ongoing or worsening signs and symptoms and testing as per Inclusion Criterion 3 above, after at least 72 hours of therapy;
5. The subject meets Inclusion Criteria 4a or 4b and has received no more than 24 hours of prior antimicrobial treatment for the current episode of CDI with oral/rectal vancomycin, IV/oral metronidazole, or oral fidaxomicin prior to Screening;
6. Female subjects of non-childbearing potential must be either surgically sterile (hysterectomy, bilateral tubal ligation, salpingectomy, and/or bilateral oophorectomy at least 26 weeks before Screening) or post-menopausal, defined as spontaneous amenorrhea for at least 2 years, with follicle-stimulating hormone in the post-menopausal range at Screening, based on the central laboratory's ranges;
7. Women of childbearing potential (ie, not post-menopausal or surgically sterilized) must have a negative urine and serum pregnancy test result before randomization. Participating women of childbearing potential must agree to use 1 highly effective method of contraception AND an acceptable barrier method (condom plus spermicide) OR 2 highly effective methods of contraception throughout the duration of the study and for 30 days following the last study drug administration. Highly effective methods of contraception that result in a low failure rate (ie, <1% per year) when used consistently and correctly include the following:

   1. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable), intrauterine device, or intrauterine hormone-releasing system for at least 12 weeks before Screening;
   2. Bilateral tubal occlusion or vasectomized partner at least 26 weeks before Screening;
   3. Sexual abstinence; NOTE: True abstinence, when in line with the preferred and usual lifestyle of the subject, is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug treatment. Periodic abstinence (eg, calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception;
8. Male subjects must agree to abstain from sperm donation and use condoms with spermicide during sexual intercourse between Screening and at least 90 days after administration of the last dose of study drug. Male subjects must ensure non pregnant female partners of childbearing potential comply with the contraception requirements in Inclusion Criterion 8.

Exclusion Criteria:

Subjects will not be enrolled in the study if they meet any of the following exclusion criteria:

1. The subject is likely to require surgical intervention (eg, subjects with fulminant CDI who fail to respond and progress to systemic toxicity, peritonitis, or toxic colonic dilatation and bowel perforation) and/or be switched to an already approved treatment regimen in the coming 48 hours due to a rapidly degrading condition;
2. The subject displays evidence of acute renal impairment with a creatinine clearance of <50 mL/min as measured by the Cockcroft Gault formula;
3. The subject is receiving hemodialysis or continuous venous hemofiltration;
4. The subject has ALT or AST serum levels >1.5 × ULN, and total bilirubin serum concentration > ULN per the testing laboratory;
5. The subject displays evidence of chronic hepatic impairment (Child-Pugh class B or C);
6. The subject is pregnant or breastfeeding;
7. The subject requires the ongoing use of anti-motility agents (eg, anti-diarrheals, anti peristaltics) or laxatives, unless approved by the Medical Monitor. Chronic and continued use of such products may be permitted during the study if bowel motility has stabilized;
8. The subject requires the ongoing use of concomitant antibiotics to treat CDI (other than study drug) (eg, oral/rectal vancomycin, IV/oral metronidazole, oral fidaxomicin) or IV immunoglobulin;
9. The subject requires the ongoing use of medications that are substrates and/or inhibitors of P glycoprotein (P-gp) or breast cancer resistance protein (BCRP). Subjects who are on such medications can be enrolled in the study if that medication can be safely stopped or replaced by another appropriate medication for the duration of the Treatment Period. Use of medications that are known P gp/BCRP substrates and/or inhibitors is permitted after completion of the Treatment Period
10. The subject has a known hypersensitivity or intolerance to DNV3837 or sorbitol;
11. The subject has a history of active hepatitis B virus or hepatitis C virus that requires ongoing therapy, or human immunodeficiency virus with the most current cluster of differentiation 4 (CD4+) <200 copies/mL;
12. The subject has participated in other clinical research studies using an investigational antibacterial or non antibacterial agent within 1 month prior to Screening;
13. The subject is unable or unwilling, in the judgment of the Investigator, to comply with the protocol; or
14. The subject is an employee of the Investigator, study site, Sponsor, or contract research organization with direct involvement in the proposed study or other studies under the direction of the Investigator, study site, or Sponsor, or a family member of the site employee or the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of diarrhea | Day 12
Treatment Success at Test of Cure | 12 days
  No relapse - Relapse is defined as a new episode of diarrhea (>3 liquid stools or UBMs [Bristol Stool Scale 6 or 7]) that results in the subject receiving antimicrobial treatment active against C. difficile. Confirmed relapse is further defined as a new episode of diarrhea (>3 liquid stools or UBMs [Bristol Stool Scale 6 or 7]) with a positive C. difficile free toxin test and the requirement of antimicrobial treatment active against C. difficile;
  * Alive;
  * No additional antimicrobial or anti-diarrheal therapies for CDI
All-Cause Mortality | Day 30
Clostridium difficile Infection attributable mortality | Day 30
Incidence of relapse at Test of Cure | 12 days
Treatment failure at Test of Cure | 12 days

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - Pinnacle Research Group, Anniston, Alabama
  - University of California (UC) Davis Medical Center, Sacramento, California
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - Infectious Disease Consultants (IDC) Clinical Research, Wichita, Kansas
  - Mercury Street Medical, Butte, Montana
  - DiGiovanna Institute for Medical Education and Research, North Massapequa, New York
  - Temple University Hospital, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Southern Star Research Institute, LLC., San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - The Medical Arts Health Research Group - Kelowna, Kelowna, British Columbia
  - Health Sciences Center, Eastern Health, Saint Johns, Newfoundland and Labrador

IPD SHARING:
Plan to Share IPD: Undecided